CLINICAL TRIAL: NCT04665401
Title: Personalizing Interventions Using Real-World Interactions: Improving Symptoms and Social Functioning in Schizophrenia With Tailored Metacognitive Therapy
Brief Title: Personalizing Interventions Using Real-World Interactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kyle S. Minor, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MERIT EAR Study
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Social Interaction; Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MERIT (Active Comparator): 24 sessions of Metacognition Reflection and Insight Therapy
  Interventions: Behavioral: Standard MERIT
- Tailored MERIT (Experimental): 24 sessions of personalized Metacognition Reflection and Insight Therapy (sessions personalized using real-world interactions)
  Interventions: Behavioral: Tailored MERIT

INTERVENTIONS:
Behavioral: Tailored MERIT — see arm description
  Arms: Tailored MERIT
Behavioral: Standard MERIT — see arm description
  Arms: Standard MERIT

SUMMARY:
Social functioning deficits are among the most disabling and difficult to treat aspects of schizophrenia. An essential component of social functioning is metacognition-a process that is profoundly disrupted in schizophrenia and represents the ability to reflect upon the mental states of oneself and others. To date, treatment efforts in schizophrenia have been hindered by barriers in accurately monitoring client's real-world social interactions. Recently, wearable technologies have evolved to provide therapists with innovative, ecologically-valid tools. The Electronically Activated Recorder is a wearable audio recorder that collects behavioral samples at pre-programmed intervals; it holds great promise as a method for yielding concrete, real-world examples of social interactions that can be used by therapists in session to enhance metacognition. Despite the immense costs of social functioning deficits, no previous studies have investigated whether functioning can be improved by integrating wearable audio recorders with psychosocial interventions.

By enhancing therapy using a wearable recording device, this proposal's primary goal is to implement a novel intervention that targets metacognitive deficits to improve social functioning. The novel intervention will be tailored to individual clients-based on the content of recorded social interactions-in a way that is not possible using traditional psychotherapy. This will allow clients and therapists to step out of the therapy room by offering a window into how clients process material in real-world interactions. In this study, a randomized controlled trial will be conducted with two schizophrenia groups receiving six months of individualized: 1) Metacognition Reflection and Insight Therapy (MERIT) alone (Standard MERIT); and 2) Tailored MERIT using wearable audio recorders. In this study, our specific aims will test feasibility, effectiveness, and acceptability of Tailored MERIT.

ELIGIBILITY:
Inclusion Criteria:

* Positive screen for metacognitive dysfunction
* Serious Mental Illness diagnosis (schizophrenia-spectrum)
* Age 18-60
* English fluency
* Currently in non-acute phase of illness

Exclusion Criteria:

* Inability to provide informed consent
* Current substance dependence
* Documented intellectual disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Global Functioning Scale: Social (GFS) | Change from baseline social functioning to social functioning after 6 months of MERIT
  10-point measure of social functioning (1 to 10, with increasing scores indicating greater social functioning)
Metacognitive Beliefs Questionnaire-Brief (MCQ-30) | Change from baseline metacognition to metacognition after 6 months of MERIT
  30 item measure of metacognition; each item is rated on a 1 to 4 scale with decreasing scores representing better metacognitive functioning.
The Positive and Negative Syndrome Scale (PANSS) | Change from baseline symptoms to symptoms after 6 months of MERIT
  30 item measure of symptoms; each item is rated 1 to 7, with greater scores representing more severe symptoms (and lower scores indicating better functioning)
EAR Adherence | Average of EAR adherence from baseline and 6 month assessment sessions
  Objective measure of how often EAR was worn; 0 (not worn) and 1 (worn) scores given at each of 48 potential time points. Total score represents frequency that the EAR is worn across all time points.
EAR Experiential Questionnaire | Average of EAR acceptability from baseline and 6 month assessment sessions
  Assessment of how acceptable wearing the EAR was and how typical days were that EAR was worn. Scores for each item range from 1 to 5 with greater scores indicating greater problems (and lower acceptability).

SECONDARY OUTCOMES:
Quality of Life Scale | Change from baseline quality of life to quality of life after 6 months of MERIT
  21 item measure of quality of life; each item is rated from 0 to 6, with greater scores indicating greater quality of life.
Metacognition Assessment Scale- Abbreviated (MAS-A) | Change from baseline metacognitive capacity to metacognitive capacity after 6 months of MERIT
  Clinician-rated measure of metacognition using a semi structured clinical interview; four areas of capacity are rated (0 to 28 on overall scale); for each, increasing scores represent greater capacity.
Short Form Health Survey (SF-36 | Change from baseline functioning to functioning after 6 months of MERIT
  36 item measure of social functioning and general health behaviors; each item on a different scale but greater scores indicate better overall functioning.
Objective Behaviors from the Electronically Activated Recorder | Baseline, 3 months into MERIT, 6 months into MERIT (MERIT completed)
  EAR coding can be implemented to rate different forms of objective behaviors; codes generated using different scales but primarily use a 0 (not present) or 1 (present) coding scheme. Greater scores typically represent presence of that which is being coded.
Scale to Assess Unawareness of Mental Disorder | Baseline, 3 months into MERIT, 6 months into MERIT (MERIT completed)
  Insight measure; three items rated on 1 to 5 scale, with increasing scores indicating poorer insight.

IPD SHARING:
Plan to Share IPD: No